CLINICAL TRIAL: NCT04976023
Title: The Effects of Using Yupingfeng Powder with Variation for the Treatment of Allergic Rhinitis(AR):a Randomized Controlled Trial
Brief Title: The Effects of Using Yupingfeng Powder with Variation for the Treatment of Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Lin Zhixiu (Other)
Responsible Party: Sponsor-Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A.Rhinitis study
Record Dates: First submitted 2021-06-10; First posted 2021-07-26 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Yupingfeng Powder variation
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Active Comparator): 14.55g of Yupingfeng Powder granules twice daily for 8 weeks
  Interventions: Drug: Yupingfeng Powder granules
- Placebo Arm (Placebo Comparator): 14.55g of placebo granules twice daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Yupingfeng Powder granules — 14.5 5 g twice daily for 8 weeks
  Other Names: Yupingfeng Powder with variation
  Arms: Active Arm
Other: Placebo — 14.5 5 g twice daily for 8 weeks
  Other Names: Placebo granules
  Arms: Placebo Arm

SUMMARY:
Allergic rhinitis (AR) is an IgE mediated chronic inflammatory disease of the upper airways characterized by symptoms of sneezing, rhinorrhea, nasal itching, and nasal obstruction . However, not only this disease is difficult to cure, but also its relapse rate is high, therefore exerting a certain impact on their daily life, work and study. Nowadays, the main treatment for allergic rhinitis is the use of western medicine, such as steroids and antihistamines. However, many clinical studies have found that the curative effect of western medicine is often not ideal.

Allergic rhinitis belongs to the category of "Rhinitis" in Chinese medicine. From the perspective of Chinese medicine, this disease is resulted from the deficiency of Qi and Yang Qi in the lungs, spleen and kidneys. Therefore, according to Chinese medicine theory, tonifying lung and spleen qi is the treatment principle for AR patients. Among different Chinese herbal formulae for AR, Yupingfeng san is commonly used for allergic diseases and in AR patients, due to its warm nature and able to improve the functions of the lungs and spleen. Yupingfeng san can improve symptoms and quality of life, as well as decrease the levels of interleukin and IgE in AR patients. This study will use Yupingfeng Powder with variation to evaluate its effectiveness and safety in treating AR. Hence, this study would be able to provide evidence on the efficacy and safety of Yupingfeng Powder with variation for AR.

DETAILED DESCRIPTION:
Rhinitis is broadly defined as inflammation of the nasal mucosa. It is a common disorder that affects up to 40% of the population. Allergic rhinitis (AR) is the most common type of chronic rhinitis, affecting 10-20% of the population, and evidence suggests that the prevalence of the disorder is increasing. AR is a very common clinical disease that can occur at any age. Severe allergic rhinitis has been associated with significant impairments in quality of life, sleep and work performance.

Allergic rhinitis is a complex immune and inflammatory disease. Its pathogenesis has not yet been fully known, and there is no clear way to cure. It is an IgE-mediated chronic inflammatory disease of the upper airways characterized by symptoms of sneezing, rhinorrhea, nasal itching, and nasal obstruction, and cytokines such as IL-17 and IL-10 play an essential role in mediating allergic inflammation. Nowadays, the main treatment for allergic rhinitis is the use of western medicine, such as steroids and antihistamines. However, many clinical studies have found that the curative effect of western medicine is often not ideal.

Chinese herbal medicine (CHM) is a well tolerated choice for AR patients seeking complementary and alternative therapies to reduce AR symptoms. In recent years, studies have found that Yupingfeng Powder not only has few side effects (feeling of abdominal distension or increased in acne are reported), it can al so increase anti allergic ability and improve body's resistance, thus showing the advantages of oral Chinese medicine in the treatment of AR. Accordingly, CHM may influence the gastrointestinal system, including the intestinal mucosa and gut microbiota, the latter of which is essential for health and closely linked to diseases. A few systematic reviews and studies indicate that certain probiotics are beneficial for patients with AR.

In this study, fifty-eight eligible subjects will be recruited from Paediatric out-patient clinic and community, and randomly assigned to receive orally Yupingfeng Powder with variation or placebo twice a day for 8 weeks, with follow-up for another 8 weeks after stopping the treatment to observe the duration of efficacy and to explore the mechanism of Yupingfeng Powder in treating AR with respect to the immune response and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age d above 5;
* Subjects with deficiency of lung and spleen Qi;
* At least 2 or more allergic symptoms rhinorrhea , sneezing , nasal obstruction and nasal itching for a cumulative period greater than 1 hour per day. These symptoms may be accompanied by itchy and red eyes and tears;
* Positive srum IgE test;
* Voluntary written consent.

Exclusion Criteria:

* Known chronic disease such as asthma, rhinosinusitis, nasal polyposis;
* Known severe medical conditions, such as cardiovascular, liver or renal dysfunction, diabetes mellitus, cancers, cerebrovascular diseases, blood system diseases;
* Concomitant steroid, nonsteroidal anti inflammatory drugs (NSAIDs), anticoagulant, and immunotherapy within past month;
* Impaired hematological profile and liver / renal function;
* Known alcohol and / or drug abuse;
* Known allergic history to any Chinese herbal medicines;
* Subjects who are pregnant or lactating.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
The change in the Total Nasal Symptom Score (TNSS) | Week 8
  The TNSS evaluates 4 nasal symptoms ( rhinorrhea, sneezing, nasal obstruction and nasal itching) which will be self assessed by subjects using a four point scale, with low scores indicating less severe nasal symptoms
The changes in quality of life by using The changes in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | week 8
  The lower the score the higher the quality of life

SECONDARY OUTCOMES:
The change in the Total Nasal Symptom Score (TNSS) | week 4, week 12 and week 16
  The TNSS evaluates 4 nasal symptoms ( rhinorrhea, sneezing, nasal obstruction and nasal itching) which will be self assessed by subjects using a four point scale, with low scores indicating less severe nasal symptoms
The changes in frequency of AR episodes and their severity on visual analog scale (VAS) | week 4, week 8, week 12 and week 16
  The VAS ranges from 0 (nasal symptom free) to 10 (nasal symptom extremely bothersome) to assess the severity of nasal symptom disturbance
The changes in quality of life by using The changes in the Paediatric Allergic Disease Quality of Life Questionnaire (PADQLQ) | week 4, week 8, week 12 and week 16
  The lower the score the higher the quality of life
The changes in quality of life by using The changes in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | week 4, week 12 and week 16
  The lower the score the higher the quality of life
The changes in the serum levels of specific IgE | week 8 and week 12
  The serum levels of cytokines and IgE will be tested. The higher the value, the more severity of the symptoms.
The changes in the serum levels of cytokines (IL-10 and IL-17) | week 8 and week 12
  Serum responses will correlate with the nasal symptoms scores.
The changes in the gut microbiota composition in stools | week 8
  The composition of gut microbiota will be tested to observe the influence of Chinese. Gut microbiome compositions will be characterised by shotgun sequencing total DNA extracted from stools.
Adverse events related to study treatment | During study for 16 weeks
  All adverse events that are related to the study treatment will be captured for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine, The Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin ZX, Ho TM, Xian YF, Chan KL, Xu QQ, Lo CW, Wu JCY, Hon KL, Leung SB, Chia CP, Sum CH, Chow TY, Cheong PK, Ching JYL, Zhang H, Leung KC, Lin WL. Exploring the efficacy and safety of Yu-Ping-Feng powder with variation against allergic rhinitis: a randomized, double-blind, placebo-controlled trial. Chin Med. 2025 May 26;20(1):70. doi: 10.1186/s13020-025-01120-2. PMID 40420199
- [Derived] Cheong PK, Ho TM, Chan KL, Lo CW, Leung SB, Hon KL, Leung KC, Siu THC, Song TH, Zhang H, Ching JYL, Chow TY, Sum CH, Chia CP, Lin ZX. The efficacy and safety of Yupingfeng Powder with variation in the treatment of allergic rhinitis: Study protocol for a randomized, double-blind, placebo-controlled trial. Front Pharmacol. 2022 Dec 16;13:1058176. doi: 10.3389/fphar.2022.1058176. eCollection 2022. PMID 36588672